CLINICAL TRIAL: NCT01963624
Title: Multicenter Prospective Study to Evaluate the Value of Combined Elastography and Color Doppler Ultrasonography for Breast Screening With Ultrasound
Brief Title: Combined Elastography and Color Doppler Ultrasonography for Breast Screening With Ultrasound
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: Elasto-Doppler Ultrasonography
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast; Screening; Ultrasound; Elastography; Doppler ultrasonography
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast masses detected with screening US: Those assessed with conventional B-mode US alone and those assessed with combined elastography and color doppler ultrasonography along with B-mode US.
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Comparison of B-mode US alone and combined use of elasto-doppler US along with B-mode US.
  Other Names: Aixplorer system (SuperSonic Imagine, France); EUB-series/HV-ASCENDUS (Hitachi Medical, Japan)

SUMMARY:
The investigators hypothesis is that the combined use of elastography and color doppler ultrasonography can increase positive-predictive value of breast screening with ultrasound.

DETAILED DESCRIPTION:
* Asymptomatic women who undergo breast screening with ultrasound and has breast masses of Breast Imaging Reporting and Data System (BI-RADS) category 3 or higher will be examined with conventional B-mode US as well as combined elasto-doppler US by breast radiologists.
* The likelihood of malignancy and BI-RADS category of the breast masses are assessed for each dataset of B-mode US alone and B-mode US with elasto-doppler US, respectively.
* Reference standard: Biopsy or 1 year of follow-up examination.
* The positive-predictive value, sensitivity, specificity, and diagnostic accuracy (assessed by the area under the receiver operating characteristic curve) are evaluated and compared between B-mode US alone and B-mode US with elasto-doppler US.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 years or older screened with breast ultrasound without specific symptoms
* Women who underwent mammography within 3 months which showed no abnormality except for dense breast
* Women who had at least one breast mass of BI-RADS category 3 or higher.

Exclusion Criteria:

* Women with breast implants
* Women who are unwilling or unable to provide informed consent
* Lesions larger than 3 cm
* Lesions that are previously noted and followed-up in the same hospital

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population will consist of asymptomatic women who visit the hospital for breast screening.
  The sites are located in 4 cities of South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 1241 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of breast screening with US | 1 year after enrollment
  Stability for 1 year of follow-up is needed for the confirmation of benign lesions if they do not undergo biopsy.

SECONDARY OUTCOMES:
Sensitivity | 1 year after enrollment
  Stability for 1 year of follow-up is needed for the confirmation of benign lesions if they do not undergo biopsy.
Specificity | 1 year after enrollment
  Stability for 1 year of follow-up is needed for the confirmation of benign lesions if they do not undergo biopsy.
Diagnostic accuracy | 1 year after enrollment
  Stability for 1 year of follow-up is needed for the confirmation of benign lesions if they do not undergo biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (10):
- South Korea (10):
  - Dongnam Inst. of Radiological and Medical Sciences, Busan
  - Gyeongsang National University Hospital, Jinju
  - CHA Bundang Medical Center, School of Medicine, CHA University, Seongnam-si
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul
  - Hanyang University Medical Center, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Seoul Metroplitan Government-Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital Healthcare System Gangnam Center, Seoul
  - Seoul National University Hospital, Seoul